CLINICAL TRIAL: NCT02987660
Title: Comparison of Topography Guided LASIK With WaveLight® EX500 to SMILE With Zeiss VisuMax
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: management decision; non patient safety related reason
Sponsor: Alcon, a Novartis Company (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RFL605-P001
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Results first posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2018-07

CONDITIONS: Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LASIK with EX500 (Experimental): Topography Guided LASIK with WaveLight EX500 excimer laser system in bilateral surgery
  Interventions: Procedure: Topography Guided LASIK; Device: WaveLight EX500 Excimer Laser System
- SMILE with VisuMax (Active Comparator): Small incision lenticular extraction (SMILE) with VisuMax laser in bilateral surgery
  Interventions: Procedure: Small Incision Lenticular Extraction; Device: VisuMax Surgical Laser

INTERVENTIONS:
Procedure: Topography Guided LASIK — Corneal surgery for refractive error correction
  Arms: LASIK with EX500
Procedure: Small Incision Lenticular Extraction — Refractive surgical procedure for the correction of myopia with or without astigmatism
  Other Names: SMILE
  Arms: SMILE with VisuMax
Device: WaveLight EX500 Excimer Laser System — As used for corneal stroma ablation (refractive error correction). The treatment is intended to last the subject's lifetime.
  Arms: LASIK with EX500
Device: VisuMax Surgical Laser — As used for lenticule creation/removal (refractive error correction). The treatment is intended to last the subject's lifetime.
  Arms: SMILE with VisuMax

SUMMARY:
The purpose of this study is to compare Topography Guided Laser In Situ Keratomileusis (LASIK) corneal surgery to Small Incision Lenticule Extraction (SMILE) corneal surgery for the treatment of myopia with astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* Subjects in Singapore must be 21 years of age or older and subjects in Korea must be upon completion of 19 years of age or older due to local regulations;
* Able to comprehend and sign an informed consent form;
* Willing and able to complete all postoperative visits;
* Myopia requiring (a) refractive error correction of -0.5 to -8.0 D optical infinity adjusted manifest refraction sphere with (b) astigmatism correction of -0.75 to -5.0 D manifest refraction cylinder and (c) at least 0.75 D of corneal astigmatism.
* Intended treatment targeted for emmetropia;
* Preoperative best-corrected visual acuity (BCVA) of 0 logMAR or better;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Pregnant or lactating, current or planned, during the course of the study;
* Dry eye;
* Corneal disease;
* Diagnosis of advanced glaucoma;
* Uncontrolled diabetes;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2017-07-26 (Actual); Study Completion 2017-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcon, A Novartis Division, Study Director — Alcon, A Novartis Division
Locations (1):
- Alcon Investigative Site, Paris, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 1 study center located in France.
Pre-assignment Details: Of the 21 enrolled, 1 subject was exited as a screen failure prior to randomization. This reporting group includes all randomized subjects (20).
Groups:
- LASIK: Topography Guided LASIK with WaveLight EX500 excimer laser system in bilateral surgery
- SMILE: Small incision lenticular extraction (SMILE) with VisuMax laser in bilateral surgery
Period: Overall Study
Arm/Group | LASIK | SMILE
Started (All randomized subjects) | 10 | 10
Completed | 0 | 0
Not Completed | 10 | 10
Not completed — Study terminated by sponsor | 10 | 10

BASELINE CHARACTERISTICS:
Population: This analysis population includes all eyes of randomized subjects for whom the treatment was initiated (Intent to treat Analysis Set) (ITT).
Groups:
- Total: Total of all reporting groups
Arm/Group | LASIK | SMILE | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 10 | 10 | 20
  ≥ 65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With Manifest Refraction Cylinder Less Than or Equal to 0.5 Diopter (D) at 3 Months
Description: Manifest refraction cylinder was measured monocularly (each eye separately) at 3 or 4 meters (m) under photopic lighting conditions using a phoropter and Early Treatment Diabetic Retinopathy Study (ETDRS) chart. The manifest refraction at 4 m or 3 m was adjusted for optical infinity by adding -0.25 D to the sphere value. Both eyes contributed to the analysis. Since the study was terminated early, inferential statistics could not be completed.
Time Frame: Month 3
Population: ITT with non-missing data
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | LASIK | SMILE
Number analyzed (Participants) | 5 | 7
Number analyzed (Eyes) | 10 | 14
percentage of eyes | 60 [26.2 to 87.8] | 100.0 [76.8 to 100.0]

2. Secondary Outcome: Mean Manifest Refraction Cylinder at 3 Months
Description: Manifest refraction cylinder was measured monocularly at 3 or 4 meters under photopic lighting conditions using a phoropter and ETDRS chart. The manifest refraction at 4 m or 3 m was adjusted for optical infinity by adding -0.25 D to the sphere value. Both eyes contributed to the analysis. Since the study was terminated early, inferential statistics could not be completed.
Time Frame: Month 3
Population: ITT with non-missing data
Measure: Mean (Standard Deviation); unit: Diopters
Units Other Than Participants: Eyes
Arm/Group | LASIK | SMILE
Number analyzed (Participants) | 5 | 7
Number analyzed (Eyes) | 10 | 14
Diopters | -0.575 (0.4091) | -0.232 (0.1539)

3. Secondary Outcome: Mean Uncorrected Visual Acuity (UCVA) at 3 Months
Description: Uncorrected (without spectacles or other visual corrective devices) Visual Acuity (UCVA) testing was conducted monocularly in photopic conditions without glare at 3 or 4 meters. Visual Acuity (VA) is measured in "logarithm of the minimum angle of resolution" (logMAR). A lower logMAR value indicates better visual acuity. The Precision Vision illuminator cabinets and ETDRS charts were used. For subjects who could not read English letters, a numerical, Tumbling E logMAR chart was used. Since the study was terminated early, inferential statistics could not be completed.
Time Frame: Month 3
Population: ITT with non-missing data
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | LASIK | SMILE
Number analyzed (Participants) | 5 | 7
Number analyzed (Eyes) | 10 | 14
logMAR | -0.100 (0.1360) | -0.164 (0.0769)

ADVERSE EVENTS:
Time Frame: Surgery through study completion, an average of 3 months, per the early termination criteria.
Description: An adverse event (AE) is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users, or other persons, whether or not related to the investigational medical device. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol.
Groups:
- LASIK: Subjects exposed to topography guided LASIK with WaveLight EX500 excimer laser system in bilateral surgery
- SMILE: Subjects exposed to SMILE with VisuMax laser in bilateral surgery
Arm/Group | LASIK | SMILE
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2017-03-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT02987660/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT02987660/SAP_001.pdf